CLINICAL TRIAL: NCT04235270
Title: Single-center, Open-label, Single-dose, 2-period, Randomized, Crossover Phase 1 Study to Demonstrate Bioequivalence of Tadalafil Administered as a Fixed Dose Combination Formulation of Macitentan/Tadalafil (10 mg/40 mg) and as the Free Combination of 10 mg Macitentan (Opsumit) and 40 mg Tadalafil (Adcirca), and to Assess the Effect of Food on the Pharmacokinetics of the Fixed Dose Formulation of Macitentan/Tadalafil (10 mg/40 mg) in Healthy Adult Participants
Brief Title: A Study of Macitentan and Tadalafil as a Fixed Dose Combination and the Free Combination in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CR108735; 67896062PAH1006 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2020-01-16; First posted 2020-01-21 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Healthy
MeSH Terms: interventions — Tadalafil; macitentan

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 (Bioequivalence Part) (Experimental): Participants will receive Treatment A (single oral dose of an fixed dose combination [FDC] of macitentan/tadalafil [10 milligram [mg]/40 mg] in fasted conditions [test]) or Treatment B (single oral dose of a free combination of 10 mg macitentan and 40 mg tadalafil in fasted conditions [reference]) on Day 1 of Treatment Period 1 followed by Treatment B or Treatment A on Day 1 of Treatment Period 2. Study drug intake in subsequent treatment periods will be separated by a washout period of at least 10 days.
  Interventions: Combination Product: FDC of Macitentan and Tadalafil; Drug: Macitentan; Drug: Tadalafil
- Group 2 (Food-effect Part) (Experimental): Participants will receive Treatment C (single oral dose of an FDC of macitentan/tadalafil [10 mg/40 mg] in fed conditions [test]) or Treatment D (single oral dose of an FDC of macitentan/tadalafil (10 mg/40 mg) in fasted conditions [reference]) on Day 1 of Treatment Period 1 followed by Treatment D or Treatment C on Day 1 of Treatment Period 2. Study drug intake in subsequent treatment periods will be separated by a washout period of at least 10 days.
  Interventions: Combination Product: FDC of Macitentan and Tadalafil; Drug: Macitentan; Drug: Tadalafil

INTERVENTIONS:
Combination Product: FDC of Macitentan and Tadalafil — Fixed dose combination (FDC) of 1 film-coated tablet containing 10 mg of macitentan and 40 mg of tadalafil will be administered orally.
Drug: Macitentan — Macitentan 10 mg tablet will be administered orally as free combination.
  Other Names: Opsumit
Drug: Tadalafil — Tadalafil 40 mg tablet will be administered orally as free combination.
  Other Names: Adcirca

SUMMARY:
The purpose of this study is to demonstrate bioequivalence on the primary pharmacokinetic (PK) parameters of tadalafil administered as an fixed dose combination (FDC) (test) of macitentan/tadalafil (10 milligram [mg]/40 mg) and coadministered as a free combination (reference) of 10 mg macitentan (Opsumit) and 40 mg Canada-sourced tadalafil (Adcirca) in fasted conditions in healthy adult participants (Group 1) and to evaluate the effect of food on the primary PK parameters of macitentan and tadalafil administered as an FDC of macitentan/tadalafil (10 mg/40 mg) in healthy adult participants (Group 2).

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI; weight [kilogram]/height^2 [m^2]) between 18.5 and 30.0 kilogram per meter square (kg/m^2), inclusive, and body weight not less than 50.0 kg at screening
* Healthy on the basis of physical examination, and medical and surgical history, performed at screening. If there are abnormalities, the participant may be included only if the investigator judges the abnormalities to be not clinically significant. This determination must be recorded in the participant's source documents and initialed by the investigator
* Healthy on the basis of clinical laboratory tests performed at screening. If the results of hematology, coagulation, or biochemistry assessments are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant. This determination must be recorded in the participant's source documents and initialed by the investigator
* Systolic blood pressure (SBP) between 100 and 145 millimeter of Mercury (mmHg), diastolic blood pressure (DBP) between 50 and 90 mmHg, and pulse rate between 45 and 99 beats per minute (bpm; inclusive), preferably measured on the right arm, after the participant is supine for at least 5 minutes, at screening
* 12-lead electrocardiogram (ECG) without clinically relevant abnormalities, at the discretion of the investigator, measured after the participant is supine for at least 5 minutes, at screening

Exclusion Criteria:

* Female participant who is breastfeeding at screening and plans to breastfeed throughout the study
* Known allergy, hypersensitivity, or intolerance to any active substance or drugs of the same class, or any excipient of the drug formulation(s)
* History or clinical evidence of any disease and/or existence of any surgical or medical condition which might interfere with the absorption, distribution, metabolism or excretion of the study treatment(s) (appendectomy and herniotomy allowed, cholecystectomy not allowed)
* Any loss of vision in 1 or both eyes
* Known hereditary degenerative retinal disorders, including retinitis pigmentosa

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2020-01-17 (Actual); Primary Completion 2020-07-17 (Actual); Study Completion 2020-07-17 (Actual)

PRIMARY OUTCOMES:
Group 1: Maximum Observed Plasma Analyte Concentration (Cmax) of Tadalafil | Up to 216 hours post dose (Up to Day 10)
  Cmax is the maximum observed plasma analyte concentration.
Group 1: Area Under the Concentration-time Curve from Time Zero to the Last Quantifiable Concentration (AUC [0-last]) of Tadalafil | Up to 216 hours post dose (Up to Day 10)
  AUC(0-last) is the area under the plasma analyte concentration-time curve from time 0 to time of the last quantifiable (non-below quantification limit [non-BQL]) concentration, calculated by linear-linear trapezoidal summation.
Group 1: Area Under the Concentration-time Curve from Time Zero to Infinity (AUC [0-infinity]) of Tadalafil | Up to 216 hours post dose (Up to Day 10)
  AUC (0-infinity) is the area under the analyte concentration-time curve (AUC) from time zero to infinite time, calculated as the sum of AUC (0-last) and C(last)/lambda(z); wherein AUC (0-last) is area under the plasma concentration-time curve from time zero to last measurable concentration, C(last) is the last observed measurable (non-BQL) analyte concentration; and lambda(z) is apparent terminal elimination rate constant.
Group 2: Maximum Observed Plasma Analyte Concentration (Cmax) of Tadalafil and Macitentan | Up to 216 hours post dose (Up to Day 10)
  Cmax is the maximum observed plasma analyte concentration.
Group 2: Area Under the Concentration-time Curve from Time Zero to the Last Quantifiable Concentration (AUC [0-last]) of Tadalafil and Macitentan | Up to 216 hours post dose (Up to Day 10)
  AUC(0-last) is the area under the plasma analyte concentration-time curve from time 0 to time of the last quantifiable (non-below quantification limit [non-BQL]) concentration, calculated by linear-linear trapezoidal summation.
Group 2: Area Under the Concentration-time Curve from Time Zero to Infinity (AUC [0-infinity]) of Tadalafil and Macitentan | Up to 216 hours post dose (Up to Day 10)
  AUC (0-infinity) is the area under the analyte concentration-time curve (AUC) from time zero to infinite time, calculated as the sum of AUC (0-last) and C(last)/lambda(z); wherein AUC (0-last) is area under the plasma concentration-time curve from time zero to last measurable concentration, C(last) is the last observed measurable (non-BQL) analyte concentration; and lambda(z) is apparent terminal elimination rate constant.

SECONDARY OUTCOMES:
Group 1 and Group 2: Time to Reach Maximum Observed Plasma Analyte Concentration (Tmax) of Tadalafil and Macitentan | Up to 216 hours post dose (Up to Day 10)
  Tmax is the actual sampling time to reach the maximum observed plasma analyte concentration.
Group 1 and Group 2: Last Observed Measurable Plasma Analyte Concentration (Clast) of Tadalafil and Macitentan | Up to 216 hours post dose (Up to Day 10)
  Clast is the last observed measurable (non-below quantification limit [non-BQL]) plasma analyte concentration.
Group 1 and Group 2: Area Under the Plasma Analyte Concentration-time Curve from Time of 0 to 72 Hours Post Dosing (AUC[0-72h] of Tadalafil and Macitentan | Up to 72 hours post dose
  AUC (0-72h) is the area under the plasma analyte concentration-time curve from time 0 to 72 hours postdose, calculated by linear-linear trapezoidal summation.
Group 1 and Group 2: Apparent Terminal Elimination Half-life (t1/2) of Tadalafil and Macitentan | Up to 216 hours post dose (Up to Day 10)
  Apparent terminal elimination half-life is time measured for the plasma analyte concentration to decrease by 1 half to its original concentration. It is associated with the terminal slope of the semi logarithmic drug concentration-time curve, and is calculated as 0.693/lambda(z).
Group 1 and Group 2: Apparent Terminal Elimination Rate Constant (Lambda[z]) of Tadalafil and Macitentan | Up to 216 hours post dose (Up to Day 10)
  Lambda(z) is first-order elimination rate constant associated with the terminal portion of the curve, determined as the negative slope of the terminal log-linear phase of the drug concentration-time curve.
Group 1 and Group 2: Total Apparent Oral Clearance (CL/F) of Tadalafil and Macitentan | Up to 216 hours post dose (Up to Day 10)
  Total apparent oral clearance is clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Group 1 and Group 2: Apparent Volume of Distribution (Vdz/F) of Tadalafil and Macitentan | Up to 216 hours post dose (Up to Day 10)
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma analyte concentration of a drug. Apparent volume of distribution after oral dose (Vdz/F) is influenced by the fraction absorbed.
Group 1 and Group 2: Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Up to 6 weeks
  An AE is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Csonka D, Fishman V, Natarajan J, Stieltjes H, Armas D, Dishy V, Perez Ruixo JJ. Bioequivalence and food effect of a fixed-dose combination of macitentan and tadalafil: Adaptive design in the COVID-19 pandemic. Pharmacol Res Perspect. 2021 Oct;9(5):e00846. doi: 10.1002/prp2.846. PMID 34624174